CLINICAL TRIAL: NCT04467619
Title: Influence of Illusory Movements on Metabolism in Patients With Large Burns
Brief Title: Illusory Movements in Patients With Burns
Acronym: Immobile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Bohumil Bakalar MD, The Head of ITU, Prague Burn Center, 3rd Medical School, Prague, Charles University, Czech Republic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20200625
Record Dates: First submitted 2020-07-03; First posted 2020-07-13 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2023-08

CONDITIONS: Catabolic State; Burns; Illusions, Kinesthetic
Keywords: Functional Proprioceptive Stimulation; Illusory Movements; Physiotherapy; Large Burns; The Critically Ill; Catabolism
MeSH Terms: conditions — Burns; Illusions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Illusory Movements (Active Comparator): Phase 1: A patient enrolled in group A will have standard rehabilitation according to the instructions of the attending surgeon and performed by an independent physiotherapist from the start of the study (Day 1), and also FPS performed by a study nurse will take place for 30 minutes twice a day, 2 hours or more after the end of standard rehabilitation, for 14 days (Day 15).
  Phase 2: From Day 16 onwards, the patient will undergo standard rehabilitation only according to the instructions of the attending surgeon and performed by an independent physiotherapist for 14 days (Day 30).
  Interventions: Device: Functional Proprioceptive Stimulation
- Deferred Illusory Movements (Active Comparator): Phase 1: A patient enrolled in group B will have standard rehabilitation according to the instructions of the attending surgeon and performed by an independent physiotherapist, from the start of the study (Day 1) for 14 days (Day 15).
  Phase 2: Then, from Day 16 onwards, in addition to standard physiotherapy, FPS performed by a study nurse will take place for 30 minutes twice a day, 2 hours or more after the end of standard rehabilitation, for 14 days (Day 30).
  Interventions: Device: Functional Proprioceptive Stimulation

INTERVENTIONS:
Device: Functional Proprioceptive Stimulation — Functional Proprioceptive Stimulations (FPS) are applied on the musculo-tendinous junction. FPS mechanically stimulate the muscle spindles, mimicking the sensory signals - Ia fibers of functional movements. This neurosensory trick activates related sensory-motor areas allowing patients to feel natural movements. Because sensory & motor systems are interdependent, the central nervous system then reacts by initiating corresponding movements.
  Other Names: Illusory Movements; Kinesthetic Illusions

SUMMARY:
Background. Large burns are the cause of extensive skeletal muscle devastation. The possibilities of rehabilitation of such patients are very limited, which contributes to the risk of metabolic failure and long-term musculoskeletal disorders. Illusory movements are a relatively new method of physiotherapy, which through functional proprioceptive stimulation enables the integration and networking of muscle units and has a neurotrophic effect on the cerebral cortex. In our pilot study, we demonstrated that illusory movements significantly increased basal energy expenditure in extensively burned patients in a catabolic state and with healing impairment in the later stage of burn disease. However, the metabolic effects of illusory movements have not yet been studied.

Tested hypotheses. 1. The use of illusory movements is suitable for the rehabilitation of patients with burns on 20% or more of the total body surface area (TBSA) in the early phase of the burn disease. 2. The use of illusory movements in these patients attenuates the extent of muscle catabolism.

Method. Pragmatic crossover study. Twenty patients with burns on 20% or more of the body surface area will be divided into two groups. They will be rehabilitated early or delayed by illusory movements for 14 days. Among other things, the following metabolic parameters will be monitored: nitrogen balance, basal and resting energy expenditure (BMR, REE), insulin resistance (IR), myokinins levels, muscle mitochondrial function and their morphology, and ultrasound cross-sectional diameter of the rectus femoris muscle. The control group will consist of ten healthy volunteers, in whom resting energy expenditure before and after using illusory movements exercise will be measured.

DETAILED DESCRIPTION:
The goal of this project is to find out whether illusory movements are suitable for patients in the early phase of burn disease, and how they influence patients' metabolism.

We are going to test these hypotheses:

* The use of illusory movements is suitable for patients with burns of 20 % TBSA and more in the early acute phase of the burn disease.
* The use of illusory movements reduces the extent of muscle catabolism in patients with large burns.

Way of solution This is a pragmatic cross-over study in patients with burns of 20 % TBSA or more in the early acute phase of the burn disease, who are expected to be hospitalized for 35 days or more. Patients meeting the inclusion criteria will be divided into two groups, A (n = 10) and B (n = 10). Group C will consist of healthy volunteers (n = 10).

The study will start after patient's basic cardiopulmonary stabilization, which usually corresponds to days 3-5 after the injury.

Group A: Early illusory movements Phase 1: A patient enrolled in group A will have standard rehabilitation according to the instructions of the attending surgeon and performed by an independent physiotherapist from the start of the study (Day 1), and also FPS performed by a study nurse will take place for 30 minutes twice a day, 2 hours or more after the end of standard rehabilitation, for 14 days (Day 15).

Phase 2: From Day 16 onwards, the patient will undergo standard rehabilitation only according to the instructions of the attending surgeon and performed by an independent physiotherapist for 14 days (Day 30).

Group B: Deferred illusory movements Phase 1: A patient enrolled in group B will have standard rehabilitation according to the instructions of the attending surgeon and performed by an independent physiotherapist, from the start of the study (Day 1) for 14 days (Day 15).

Phase 2: Then, from Day 16 onwards, in addition to standard physiotherapy, FPS performed by a study nurse will take place for 30 minutes twice a day, 2 hours or more after the end of standard rehabilitation, for 14 days (Day 30).

Group C: Illusory movements in healthy individuals This group will consist of 10 healthy volunteers in whom REE will be measured before and after 30 minutes of FPS.

c) Medical, social and economic rationale of this study Large burns are often the cause of neuromyopathy and disability of the injured [30]. Hypercatabolism and enormous muscle loss increase the morbidity and mortality of patients, prolong treatment and greatly increase the overall cost of medical care [31]. Early rehabilitation using illusory movements could reduce the extent of muscle devastation in otherwise immobile patients and improve the effect of standard rehabilitation by maintaining functional brain maps. This should lead to an earlier return of the injured to their normal activities a improve quality of life.

In addition, if the positive effects of illusory movements are proved, there are many critically ill patients outside the burns who could benefit from this form of physiotherapy.

d) Methodology Nutrition support will be provided in accordance with European Society of Parenteral and Enteral Nutrition recommendations.

During the study, the following parameters will be measured, and the following examinations will be performed in addition to standard biochemical, haematological and imaging examinations of Group A and B:

Daily:

* Nitrogen balance;
* Resting Energy Expenditure using indirect calorimetry;

On Days 1, 15 and 30:

* Patient weight;
* APACHE II score;
* Muscle biopsy (from m. vastus lateralis);
* BMR;
* Glucose disposal using a hyperinsulinaemic euglycaemic clamp;
* Degree of insulin resistance according to Homeostasis Model Assessment;
* Muscle mitochondrial respiratory capacity and coupling with the Oxygraph-2K;
* Mitochondrial mass determination and dynamics in myocytes with MitoTracker® ;
* Plasmatic levels of myokinins ;
* Ultrasound measurement of the rectus femoris diameter measured by an independent sonographer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older;
* Consent to be included in the study;
* Burns II. - III. grade on 20 % TBSA and more;
* Admission within 72 hours of the accident;
* Expected hospital stay of 35 days or more.

Exclusion Criteria:

* Age <18 years;
* Refusal of the study in any point;
* Unlikely patient survival (Revised Baux Index> 120);
* Known primary neuromuscular diseases or spinal cord lesions;
* Limb amputation before or during the study;
* Bed rest before admission;
* Pregnancy;
* External fixator or surface metal implant on the limbs;
* Known malignancy or history of malignancy treatment in the last 5 years;
* History of HIV or AIDS;
* Concomitant treatment with systemic corticosteroids;
* Pacemaker, implanted defibrillator, or another bio-electronic device;
* Patient in prison.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Energy expenditure | 2 years
  The use of illusory movements changes energy expenditure in patients with large burns.
Anticatabolic effect | 2 years
  The use of illusory movements changes the extent of muscle catabolism in patients with large burns.

SECONDARY OUTCOMES:
Insulin resistance | 2 years
  The use of illusory movements changes the extent of insulin resistance in patients with large burns.
Mitochondrial functions | 2 years
  The use of illusory movements changes mitochondrial functions of skeletal muscle in patients with large burns.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Kralovske Vinohrady, Prague, Czechia

REFERENCES:
- [Background] Roll R, Kavounoudias A, Albert F, Legre R, Gay A, Fabre B, Roll JP. Illusory movements prevent cortical disruption caused by immobilization. Neuroimage. 2012 Aug 1;62(1):510-9. doi: 10.1016/j.neuroimage.2012.05.016. Epub 2012 May 12. PMID 22584228
- [Background] Jeschke MG, van Baar ME, Choudhry MA, Chung KK, Gibran NS, Logsetty S. Burn injury. Nat Rev Dis Primers. 2020 Feb 13;6(1):11. doi: 10.1038/s41572-020-0145-5. PMID 32054846
- [Background] Waldauf P, Jiroutkova K, Krajcova A, Puthucheary Z, Duska F. Effects of Rehabilitation Interventions on Clinical Outcomes in Critically Ill Patients: Systematic Review and Meta-Analysis of Randomized Controlled Trials. Crit Care Med. 2020 Jul;48(7):1055-1065. doi: 10.1097/CCM.0000000000004382. PMID 32345834